CLINICAL TRIAL: NCT06885723
Title: Evaluation of Different Anesthesia Methods to Reduce Pain From Intratympanic Injections: A Prospective, Randomized Clinical Trial
Brief Title: Use of Vibration Anesthesia Device in Intratympanic Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ramazan Akin, MEDİCAL DOCTOR, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Desicion No:03 Date:17.06.2020
Record Dates: First submitted 2024-12-23; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intratympanic Injections; Sudden Hearing Loss
Keywords: sensorineural hearing loss; VAD; intratympanic steroid; pain; Sudden hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss, Sensorineural; Pain

STUDY DESIGN:
Intervention Model Description: Prior to each intratimpanik steroid injection (ITS), all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient. After each ITS, pain assessment was performed using Visual Analogue Scale , Numerical Rating Scales, and Verbal Rating Scales
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1.group (Experimental): Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient. After each ITS, pain assessment was performed using Visual Analogue Scale (VAS), Numerical Rating Scales (NRS), and Verbal Rating Scales (VRS)
  Interventions: Device: Vibration Anesthesia Device (VAD)
- 2.group (Active Comparator): Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Interventions: Drug: local anesthetic cream
- 3.group (Active Comparator): Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Interventions: Drug: lidocaine spray
- 4.group (Placebo Comparator): Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Interventions: Other: saline drops

INTERVENTIONS:
Device: Vibration Anesthesia Device (VAD) — In conclusion, induction of anesthesia with VAD in patients treated with ITS provided pain palliation in a similar way to other local anesthetic techniques. Moreover, the advantage of VAD application over other anesthetic agents was that it eliminated the need to use local anesthetics that may disrupt wound healing. In addition, inducing anesthesia with VAD can be considered as an alternative method in patients allergic to drugs. Our study will shed light on different techniques such as the application of ventilation tube in anesthesia with VAD.
  Arms: 1.group
Drug: local anesthetic cream — Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Arms: 2.group
Drug: lidocaine spray — Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Arms: 3.group
Other: saline drops — Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. The order of administration was determined for each patient using the randomization software (random.org/lists/). For the fifth ITS, however, the method of administration was selected by the patient.
  Arms: 4.group

SUMMARY:
SUMMARY Intratympanic injections commonly cause pain in the patients. Intratympanic steroid injection (ITS) application can be performed by direct injection without anesthesia or with local anesthesia induced by lidocaine spray, lidocaine injection, topical phenol, pantocaine, EMLA cream (lidocaine+prilocaine) or vibration anesthesia device (VAD). The advantage of VAD application over other anesthetic agents was that it eliminated the need to use local anesthetics that may disrupt wound healing. In addition, inducing anesthesia with VAD can be considered as an alternative method in patients allergic to drugs.

DETAILED DESCRIPTION:
ABSTRACT In this study, we aimed to compare the efficacy of four methods including topical lidocaine spray, local anesthetic cream, vibration anesthesia device (VAD), and saline drops (control group) in the reduction of pain after intratympanic steroid injections (ITS's) and to demonstrate the effectiveness of VAD use. The prospective study included 40 patients aged 18-70 years with idiopathic sudden sensorineural hearing loss. Prior to each ITS, all the four methods including local anesthetic cream (EMLA® cream, AstraZeneca PLC), lidocaine spray (Vemcain® Spray), VAD (Blaine®, Blaine Labs, Santa Fe, USA), and saline drops (control) were administered in each patient. After each ITS, pain assessment was performed using Visual Analogue Scale (VAS), Numerical Rating Scales (NRS), and Verbal Rating Scales (VRS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years with idiopathic sudden sensorineural hearing loss

Exclusion Criteria:

* History of otologic surgery,
* Recent ototoxic drug use,
* Congenital inner ear malformation,
* History of chemoradiotherapy due to malignant neoplasia,
* Presence of acute or chronic otitis media,
* Age under 18 years, over 70 years
* History of local anesthesia allergy,
* Coagulation abnormality,
* Pregnant and lactating women,
* Hearing cases with other neurootological diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | 56 weeks
  Visual Analogue Scale (VAS). the visual analog scale (VAS) scaled between 0-10,were used.
Eleven-Point Numeric Rating Scale(NRS-11) | 56 weeks
  Eleven-Point Numeric Rating Scale (NRS-11). the numerical rating scale (NRS) scaled between 0-10 were used.
Four-Category Verbal Rating Scale(VRS-4) | 56 weeks
  Four-Category Verbal Rating Scale (VRS-4). the verbal rating scale (VRS) scaled between 0-4 were used.

CONTACTS AND LOCATIONS:
Locations (1):
- van yuzuncu yil university, Bardakçı, Yüzüncü Yıl Ünv., 65080 Tuşba/Van, Van, Turkey (Türkiye)